CLINICAL TRIAL: NCT04228380
Title: Limitations and Mortality in Intensive Care
Acronym: LIMO
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: LIMO
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inclusion: Inclusion criteria: The cohort is made up of adult patients over 65 years of age, admitted to an intensive care unit in Sweden, for other reason than postoperative care or simple monitoring.
  Interventions: Other: No intervention
- Exclusion: Exclusion criteria: Declined consent to participate.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is an observational prospective pilot-study that investigates which patient-related variables that predict a decision to limit life sustaining treatments. Some of the variables we were interested in cannot be accessed in registry data, such as frailty scale score and living at home or not. Furthermore we wanted to investigate if the variables that were independently associated with a decision to limit LST were different for critically ill patients with COVID-19 than for critically ill patients with other diagnoses in a Swedish intensive care unit during the pandemic.

DETAILED DESCRIPTION:
Previous publications have demonstrated variability in end-of-life decision-making (ELDM) for critically ill patients (1-3).

Factors commonly described as underlying the variability in ELDM in northern Europe are patient-related factors such as age, sex, the severity of illness, frailty, chronic poor health, and diagnosis (4-6). Variability in ELDM is also caused by other less readily identifiable factors, such as preferences and experiences of the attending physicians (7-8).

When the pandemic of the coronavirus disease 2019 (COVID-19) struck worldwide, intensive care units (ICUs) were put under immense pressure, and resources were strained to their limit. More than 550 million cases and 6.3 million deaths have been reported worldwide (9). In Sweden, more than 9000 patients with COVID-19 were admitted for intensive care, dramatically increasing the demand for intensive care resources (10).

At the beginning of the pandemic, this disease was primarily unknown to physicians in the ICU, and its course and plausible patient outcomes were difficult to predict. Factors that have been demonstrated to predict poor long-term outcomes in critically ill COVID-19 patients are extensively studied. In a Swedish setting, they were found to be male sex, high age, high simplified acute physiology score (SAPS 3) (11), the month of admission, and preexisting conditions such as obesity, asthma, chronic obstructive pulmonary disease, malignancy, and immune deficiency (12).

End-of-life decisions in critically ill patients with and without COVID-19 are closely associated with short-term mortality (13-14). There are surprisingly few studies on EDLM in COVID-19 patients and whether these decisions were handled differently compared to other critically ill patients during the pandemic (15-16). It could be postulated that the process of ELDM changed during the pandemic as increased demands for intensive care caused an explicit lack of resources (17).

We hypothesised that ELDM was challenging for COVID-19 patients due to several uncertainties concerning prognostication. Therefore, we stipulated that end-of-life decisions in COVID-19 patients were made for older patients with higher frailty scores than the non-COVID-19 cohort and that end-of-life decisions were postponed to later in the course of the COVID-19 disease. We also hypothesised that a more significant proportion of patients in the COVID-19 cohort died without any end-of-life decision being made before death compared to the non-COVID-19 cohort.

In this study, we primarily aimed to investigate which independent factors predicted a decision to withdraw or withhold life-sustaining treatments (LST) in critically ill patients if these decisions were based on different variables for critically ill patients with COVID-19 compared to critically ill patients with other diagnoses in a Swedish ICU. Secondly, we aimed to investigate if ELDM was made later in the course of the disease for COVID-19 patients and if a higher proportion of COVID-19 patients died without any decision to limit LST.

ELIGIBILITY:
Inclusion Criteria:

Patients over 65 years admitted to an intensive care unit for care other than simple monitoring or uncomplicated postoperative care.

Exclusion Criteria:

Declined consent to participate.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: I cohort with critically ill COVID-19 patients, 1 cohort with critically ill patients with other diagnosis than COVID-19.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Variables that independently impact decisions to limit LST ICU's. Differences between covid-19 and non-Covid-19 patients. | 2020-2025
  Impact of gender, age, frailty, comorbidities, invasive ventilation, SAPS 3, BMI, length of stay on decisions to limit LST in critical illness in Swedish ICU's.

SECONDARY OUTCOMES:
Secondary outcomes | 2020-2025
  The secondary outcome was the time from admission to the end-of-life decision and to investigate if a higher proportion of patients in the COVID-19 cohort died without a previous decision to limit life sustaining treatments. Furthermore, we aimed to investigate if mortality differed between the groups. In addition, we aimed to investigate if survival after a decision to limit LST differed between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Block, PhD, Principal Investigator — Shalgrenska Academy, Gothenburg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden